CLINICAL TRIAL: NCT06949969
Title: Alesis OSA-1 Double-Blinded Randomized Study of Obstructive Sleep Apnea Treatment Using A Patented Noncoherent Medical Light
Brief Title: Alesis OSA-1 Obstructive Sleep Apnea Treatment
Acronym: OSA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Photonica USA, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Device Feasibility
Other Study IDs: IORG0012434; IORG0012434 (Other: Space Coast Biomedical IRB)
Record Dates: First submitted 2025-04-18; First posted 2025-04-29 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Obstructive Sleep Apnea
Keywords: OSA, Sleep Apnea, Alesis OSA1, AHI, LLLT, UltraSlim
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Apnea Syndromes

STUDY DESIGN:
Intervention Model Description: The study will compare two groups, a control group which will receive a simulated 12 minute treatment that does not expose the participant to LLLT and a treatment group who will receive a 12 minute treatment using LLLT. The Alesis OSA-1 device is a branded UltraSlim Digital device that uses narrowband 635nm noncoherent light to immediately reduce fat volume. The device has three 510(k) FDA clearances (K160880, K150336, and K202361).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (4):
- Alesis OSA-1 Effectivness (Active Comparator): The treatment group of the study will receive LLLT from the previously FDA 501(k) class I approved Ultraslim device, now rebranded under the name Alesis OSA-1. N=35 participants will receive non-invasive LLLT at 635nm wavelength for 12 minutes, 2x per week, x 3 weeks.
  The Alesis OSA-2 device will be used for this arm of the study.
  Interventions: Device: OSA LLLT treatment device
- MRI Assessment (No Intervention): 5 participants from the treatment group will be randomly selected to receive to pre and post magnetic resonance imaging (MRI) on the head/neck to determine change in size or volume of soft tissue and fat within the airway/neck structures.
- PFT Assessment (No Intervention): Ten participants, 5 from the treatment group and 5 from control, will receive pre and post study pulmonary function testing (PFT) to evaluate changes in pulmonary volumes related the treatments.
- OSA-1 Control group (Placebo Comparator): A modified device utilizing a pigtail connector to bypass active treatment while allowing the cooling fans to operate for the treatment period, giving the appearance of treatment with invisible light.
  Interventions: Device: Sham Comparator

INTERVENTIONS:
Device: OSA LLLT treatment device — The Alesis OSA-1 is a LLLT that uses 635nm wavelength to stimulate the mitochondria to open cell spaces and allow oils, lipids, and fluids to drain into the body systems.
  Arms: Alesis OSA-1 Effectivness
Device: Sham Comparator — A modified device utilizing a pigtail connector to bypass active treatment while allowing the cooling fans to operate for the treatment period, giving the appearance of treatment with invisible light.
  Arms: OSA-1 Control group

SUMMARY:
The goal of randomized clinical trial is to determine if the Alesis OSA-1 low laser light therapy device can reduce apnea-hypopnea index scores and treat sleep apnea in adult participants over the age of 18 who are diagnosed with obstructive sleep apnea (OSA). The main questions it aims to answer are]:

• Does the use of the Alesis OSA-1 device reduce the number of AHI events after six treatments of 12 minutes each, 2x per week x 3 weeks, in adult OSA patients?

Researchers will compare results of 35 control group participants who will not receive treatment to a treatment group who will receive six, 12 minute, non-invasive low laser light therapy (LLLT) treatments, two per week for 3 weeks, to see if there is a reduction in the number of AHI events and size of redundant and soft tissues in adult OSA patients.

Participants will:

* Visit the clinic for assessment and instructions on using the at home sleep study system, WatchPat, and obtain baseline information
* Use the WatchPat system to record AHI events pre- and post-treatment.
* 10 randomly selected participants will receive a pre-study pulmonary functions test (PFT) and repeated post-treatment.
* 5 randomly selected participant will receive a pre-study MRI of the head/neck and repeated post treatment.
* For the treatments, the participant lie on a treatment table under a LLLT device for 12 minutes, two times per week, x 3 weeks.
* Be offered the treatment series at the conclusion of the study if they were selected for the control group.

DETAILED DESCRIPTION:
PURPOSE To evaluate the efficacy of the non-invasive Alesis Low-Level Light Therapy (LLLT) medical device in treating obstructive sleep apnea (OSA) by assessing changes in upper airway fat deposits via. Magnetic resonance imaging (MRI) after treatments; Apnea-Hypopnea Index (AHI) events; and STOP-BANG scores pre- and post-treatment; determining its potential to reduce fat and improve airway patency in adults with mild to severe OSA.

OBJECTIVES

* To evaluate changes in the size of the tongue and soft tissue structures in obese subjects diagnosed with obstructive sleep apnea (OSA).
* To assess improvements in the Apnea-Hypopnea Index (AHI) following treatment with the Alesis Airway LLT Modification Device.

STUDY DESIGN

* Type: Prospective, repeated measures, double blind, randomized controlled trial
* Participants: N = 70 for original study, N = 5-10 MRI subset, N = 35 for ethical consideration offering (See Ethics considerations)
* Sampling Method: Volunteer convenience sample
* Duration: 6 months
* Special subset A: A subset of 3-10 participants will undergo a MRI evaluation to measure submental and tongue fat size, pre- and post-treatment (Reference: Schwab, et al. 2014, Tongue fat and OSA relationship)
* Repeated Measures: Post-Treatment HST week 2, week 3

PARTICIPANTS Inclusion Criteria

* Suspicion of OSA
* STOP BANG score of 3 or greater (See STOP BANG CRITERIA)
* Age ≥ 18 years - 70
* Obese (BMI ≥ 25) Exclusion Criteria
* Beards - beard
* Central Sleep Apnea
* Inability to hold mouth open 12 minutes
* Age > 75/ < 18
* Severe comorbid conditions that may affect treatment or inability to lie flat or sit for 20 minutes (e.g., severe cardiac disease, uncontrolled diabetes)
* Contraindications to MRI (e.g., non-MRI-compatible pacemakers).
* History of recent upper airway surgery.
* Active cancer or cancer treatment completion within 1 year

DEMOGRAPHICS & COMORBIDITIES

* Demographics
* Participants Identifier Number
* Age•
* Sex
* Height
* Weight
* BMI
* Significant Comorbidities (e.g., diabetes, hypertension, cardiac disease, kidney disease, memory issues, narcolepsy)
* Comorbidities: Although not exclusion criteria, document significant medical history, including:
* Diabetes
* Hypertension
* Cardiac disease
* Kidney disease
* Memory loss or cognitive issues
* Narcolepsy
* Other relevant conditions
* Medication use contraindicated on consent

TREATMENT PROTOCOL & INTERVENTION

* Device: Alesis OSA-1
* Pre-Admission Steps
* Basic health history
* Qualitative survey for participants for anecdotal data and quotes
* STOP BANG assessment (Score of ≥ 3 )
* Consent to treat and Informed consent for study participation
* Pre-Treatment Steps
* Randomization into treatment and control groups using alternative numbering system
* Baseline height and weight
* Baseline physical measurements per tape measure on neck circumference included in the STOP BANG
* Baseline AHI Study using WatchPat device
* 3D Imaging of treatment area
* SUBSET A: 5 participants will get baseline MRI
* Measure tongue adipose, size, and structure shape
* Measure submental tissue size
* SUBSET B: 10 randomly selected participants will get pre and post

Session Details

* Duration: 12 minutes per treatment session -Facing front with mouth open
* LLLT 5 cm from face/neck
* Goggles for eye protection
* Frequency: 6 sessions over a set period (e.g., 3 weeks), 2 x week x 3 weeks
* Control group will receive light therapy with a sham connector between the control console and light/arm assembly, that operates the cooling fans with the 635nm light off in order to mimic invisible light.

Post-Treatment Steps:

* After the last treatment in week 3: Post treatment AHI test, Weight, STOP BANG score, neck circumference measurement, and qualitative questionnaire 5 questions.
* After week 3 and last week of treatment - 3D Imaging will be completed using the Vector camera system
* Qualitative data survey for participants for anecdotal data and quotes
* SUBSET A: MRI Group - MRI repeated after week 3, session 6.
* SUBSET B: PFT Group - PFTs repeated after last treatment in week 3, session 6.

Ethical Considerations

* To benefit health care and do the ethical thing for society, control group participants will be offered the intervention treatments, post-study, if results demonstrate a reduction in incidence of AHI 20% or greater.
* Control participants (Group A) that opt for the treatments post study, will utilize the home study sleep monitoring and data will be used to compare to data collected during their control group assignment.

TOOL • Home Monitoring: Participants will use the WatchPAT device to monitor AHI prior to study and repeated after 6 treatments.

MEASUREMENTS

* Pre-Treatment Assessment
* AHI Monitoring:
* Use WatchPAT devices for baseline AHI measurement.
* AHI event occurrence per hour
* Respiratory Disturbance Index data: apneas, hypopneas, respiratory effort related arousals (RERAs) per hour of sleep
* Oxygen disturbance Index data: SpO2 % drop data
* SpO2 levels via pulse oximetry: nadir/lowest, average during sleep, thresholds
* Vital signs - Heart rate average, HR variability patterns
* Total sleep time
* Latency - time to fall asleep
* REM latency - time to REM
* Sleep stage data - estimate
* Snoring intensity
* Body position
* Cheyne-stokes respirations for Central Sleep Apnea
* Movement
* Peripheral arterial tone (sympathetic responses and events
* MRI Measurements on 10 randomized participants:
* Post-Treatment Assessment
* AHI Monitoring:
* Repeat AHI measurement with WatchPAT system after the completion of all treatment sessions.
* MRI Measurements on 5-10 randomized participants:
* Repeat MRI to evaluate airway size, volume, and structure/changes

DATA ANALYSIS

* Analysis Methods:
* Compare pre- and post-treatment AHI values using paired t-tests or Wilcoxon signed-rank tests as appropriate.
* Analyze changes in MRI measurements using repeated measures ANOVA or mixed-model analysis.
* Correlation between fat loss and reduction in AHI events, STOP BANG using Pearson's Correlation Coefficient

EXPECTED OUTCOMES

* Identification of correlations between treatments and changes in the volume or tongue and submental tissue volume
* Evaluation of the effectiveness of the Alesis OSA1 treatment in reducing AHI in participants with OSA.

ETHICAL CONSIDERATIONS

* Obtain informed consent from all participants.
* Ensure confidentiality and data protection throughout the study.
* Offer post-treatment procedures to control group participants if results demonstrate 20% or greater reduction in AHI events

CONCLUSION

• This study aims to provide insights into the effects of non-invasive LLLT airway modification treatment on OSA, enhancing understanding of the relationship between soft tissue structures and apnea severity in obese individuals.

ELIGIBILITY:
Inclusion Criteria:

* Suspicion of OSA, known diagnosis of OSA, STOP BANG score of 3 or greater, BMI >/= 25

Exclusion Criteria:

* Beard or facial hair, diagnosis of central sleep apnea, inability to hold mouth open 12 minutes, Age less than 18 years old, • Severe comorbid conditions that may affect treatment or inability to lie flat or sit for 20 minutes (e.g., severe cardiac disease, uncontrolled diabetes); Contraindications to MRI (e.g., non-MRI-compatible pacemakers); History of recent upper airway surgery; Active cancer or cancer treatment completion within 1 year; Contraindications to LLLT such as systemic lupus erythematosis (SLE); Photosensitivity; Pregnancy; Renal disease; Facial fillers within 3 months; Diabetes medications (light sensitivity) Sulfonylurea medications, Metformin, Sitagliptin; Liver disease; Autoimmune disorders; Albinism; Antibiotic therapy-Tetracyclines, Fluoroquinolones (ciprofloxacin, ofloxacin, levofloxacin); Sulfonamides, Tricyclic antidepressants.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
AHI Events | From enrollment until the end of treatment at 3 weeks.
  Apnea-hypoapnea events will be documented on the at home OSA sleep study (WatchPat) device. The number of AHI events occurring pre and post treatment will be evaulated for improvement;

SECONDARY OUTCOMES:
Fat and tissue volume reduction | From enrollment to the end of treatment at 3 weeks
  Pre and post treatment MRI measurements of fat and tissue volume in the head and neck region will be compared to evaluate efficacy of the Alesis OSA-1 device to treat OSA.
Pulmonary Functions Volumes | From enrollment to end of treatment in 3 weeks
  Pre and post treatment pulmonary function studies will be compared to evaluate efficacy of the Alesis OSA-1 device to impact respiratory volumes which are reduced in OSA.

CONTACTS AND LOCATIONS:
Overall Officials: Joaquin Hechavarria, MD, Principal Investigator — JD Medical Group, LLC
Locations (2):
- United States (2):
  - JD Medical Group, LLC, Miami, Florida
  - Bioresearch Institute, Llc., Miramar, Florida

IPD SHARING:
Plan to Share IPD: Yes
Sleep study reports, Pre and post treatment MRI tissue measurements, PFT pre and post treatment volumes
Supporting Information: Study Protocol, ICF, CSR
Time Frame: The data will be available starting three months after after the study completion date and for one full year (end date).
Access Criteria: Researchers conducting similar or related studies can request the information by contacting the primary study contract in email or writing. They will receive a de-identified excel file that is password protected.
URL: https://photonicausa.com/research.php

REFERENCES:
- [Background] Medical Advisory Secretariat. Polysomnography in patients with obstructive sleep apnea: an evidence-based analysis. Ont Health Technol Assess Ser. 2006;6(13):1-38. Epub 2006 Jun 1. PMID 23074483
- [Background] Sutherland K, Lowth AB, Antic N, Carney AS, Catcheside PG, Chai-Coetzer CL, Chia M, Hodge JC, Jones A, Kaambwa B, Lewis R, MacKay S, McEvoy RD, Ooi EH, Pinczel AJ, McArdle N, Rees G, Singh B, Stow N, Weaver EM, Woodman RJ, Woods CM, Yeo A, Cistulli PA. Volumetric magnetic resonance imaging analysis of multilevel upper airway surgery effects on pharyngeal structure. Sleep. 2021 Dec 10;44(12):zsab183. doi: 10.1093/sleep/zsab183. PMID 34283220
- [Background] Wang SH, Keenan BT, Wiemken A, Zang Y, Staley B, Sarwer DB, Torigian DA, Williams N, Pack AI, Schwab RJ. Effect of Weight Loss on Upper Airway Anatomy and the Apnea-Hypopnea Index. The Importance of Tongue Fat. Am J Respir Crit Care Med. 2020 Mar 15;201(6):718-727. doi: 10.1164/rccm.201903-0692OC. PMID 31918559
- [Background] Orestes MI, Tuchayi SM, Wang Y, Farinelli W, Arkun K, Anderson RR, Thomas R, Garibyan L. Safety and feasibility of selective tongue fat reduction with injected ice-slurry. Laryngoscope Investig Otolaryngol. 2022 Sep 9;7(5):1675-1680. doi: 10.1002/lio2.902. eCollection 2022 Oct. PMID 36258870
- [Background] Kirsch DB. Obstructive Sleep Apnea. Continuum (Minneap Minn). 2020 Aug;26(4):908-928. doi: 10.1212/CON.0000000000000885. PMID 32756228
- [Background] Guo J, Xiao Y. New Metrics from Polysomnography: Precision Medicine for OSA Interventions. Nat Sci Sleep. 2023 Mar 9;15:69-77. doi: 10.2147/NSS.S400048. eCollection 2023. PMID 36923968
- [Background] Kennedy J, Verne S, Griffith R, Falto-Aizpurua L, Nouri K. Non-invasive subcutaneous fat reduction: a review. J Eur Acad Dermatol Venereol. 2015 Sep;29(9):1679-88. doi: 10.1111/jdv.12994. Epub 2015 Feb 9. PMID 25664493
- [Background] Moon IJ, Choi JW, Jung CJ, Kim S, Park E, Won CH. Efficacy and safety of a novel combined 1060-nm and 635-nm laser device for non-invasive reduction of abdominal and submental fat. Lasers Med Sci. 2022 Feb;37(1):505-512. doi: 10.1007/s10103-021-03288-z. Epub 2021 Apr 2. PMID 33797649
- [Background] Caruso-Davis MK, Guillot TS, Podichetty VK, Mashtalir N, Dhurandhar NV, Dubuisson O, Yu Y, Greenway FL. Efficacy of low-level laser therapy for body contouring and spot fat reduction. Obes Surg. 2011 Jun;21(6):722-9. doi: 10.1007/s11695-010-0126-y. PMID 20393809
- [Background] Avci P, Nyame TT, Gupta GK, Sadasivam M, Hamblin MR. Low-level laser therapy for fat layer reduction: a comprehensive review. Lasers Surg Med. 2013 Aug;45(6):349-57. doi: 10.1002/lsm.22153. Epub 2013 Jun 7. PMID 23749426
- See also: Clinical trial for LLLT in body contouring and fat reduction — https://clinicaltrials.gov/expert-search?term=NCT02867150
- See also: 510K clearance for body contouring, fat reduction, inflammation, and skin tightening. Ultraslim rebranded as Alesis OSA-1 — https://www.accessdata.fda.gov/scripts/cdrh/cfdocs/cfPMN/pmn.cfm?ID=K202361